CLINICAL TRIAL: NCT05825378
Title: The Effect of Intercostal Nerve Block With Dexamethasone and Ropivacaine on Rebound Pain After Thoracoscopic Surgery: a Randomized, Double-blind, Controlled Study
Brief Title: The Effect of Intercostal Nerve Block With Dexamethasone and Ropivacaine on Rebound Pain After Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director of Anesthesiology Department, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230411
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Rebound Pain; Dexamethasone; Intercostal Nerve Block; Thoracoscopic Surgery
MeSH Terms: interventions — Dexamethasone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group dexamethasone (Experimental): Dexamethasone 8mg+0.375% ropivacaine
  Interventions: Drug: Dexamethasone 8mg+0.375% ropivacaine
- group control (Sham Comparator): 0.375% ropivacaine
  Interventions: Drug: 0.375% ropivacaine

INTERVENTIONS:
Drug: Dexamethasone 8mg+0.375% ropivacaine — Ultrasound-guided intercostal nerve block was performed on the surgical side, and 3 to 5ml of a mixture of 0.375% ropivacaine and 8 mg dexamethasone was injected at each point
  Arms: group dexamethasone
Drug: 0.375% ropivacaine — Ultrasound-guided intercostal nerve block was performed on the surgical side, and 3 to 5ml 0.375% ropivacaine was injected at each point
  Arms: group control

SUMMARY:
Regional nerve block is one of the commonly used methods for postoperative analgesia after thoracoscopic surgery. Recent studies have found that rebound pain may occur after regional block, which is defined as acute postoperative pain that occurs after the resolution of sensory block related to regional anesthesia, and seriously affects the quality of postoperative recovery of patients. There is evidence that rebound tenderness is associated with local anesthetic toxicity and proinflammatory effects. The aim of this study was to investigate the effect of dexamethasone on rebound pain after a single intercostal nerve block in patients undergoing thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective thoracoscopic surgery Age > 18 years old ASA ⅰ-ⅲ Informed consent was signed

Exclusion Criteria:

* Patients with aoagulation disorders Patients with allergy to local anesthetics Patients with severe cardiopulmonary diseases Patients had systemic steroid use Patients with chronic pain Patients with uncontrolled diabetes and mental disorders History of drug abuse; Body Mass Index more than 35 kg.m-2 Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-08-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of rebound pain after the disappearance of nerve block effect | 8 hours after the nerve block
  NRS < 3 in PACU and NRS > 7 after the disappearance of nerve block effect

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No